CLINICAL TRIAL: NCT03805633
Title: A Suspected Association Between Sarcoidosis and Development of Diabetes Mellitus
Status: Withdrawn | Type: Observational
Why Stopped: Person working on the trial left
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Fernando Ovalle, Medical Doctor, Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300000289
Record Dates: First submitted 2018-01-22; First posted 2019-01-16 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Sarcoidosis; Diabetes Mellitus
MeSH Terms: conditions — Sarcoidosis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sarcoidosis Patients: Patients referred to UAB Pulmonology who are diagnosed with sarcoidosis.
  Interventions: Diagnostic Test: Venous blood sample; Diagnostic Test: Ultrasound of pancreas
- Diabetes Patients: Patients followed by UAB Endocrinology with diabetes mellitus.
  Interventions: Diagnostic Test: Venous blood sample; Diagnostic Test: Ultrasound of pancreas
- Sarcoidosis and Diabetes patients: Patients followed by UAB Pulmonary and/or UAB Endocrinology with both sarcoidosis and diabetes mellitus.
  Interventions: Diagnostic Test: Venous blood sample; Diagnostic Test: Ultrasound of pancreas

INTERVENTIONS:
Diagnostic Test: Venous blood sample — Venous blood samples will be obtained for hemoglobin A1c, C peptide, insulin level, and 2-hour fasting glucose tolerance test.
Diagnostic Test: Ultrasound of pancreas — Ultrasound of pancreas will be obtained on all study participants.

SUMMARY:
The purpose of the study is to determine the characteristics of patients with diabetes and sarcoidosis and to compare them with those of patients with diabetes and no sarcoidosis. The investigators will approach these aims by measuring hemoglobin A1c, C peptide, insulin levels, and 2-hour glucose tolerance test results on the study population as well as collecting clinical data from records. Three groups of patients will be identified from pulmonary and endocrinology clinics at the University of Alabama at Birmingham. The first group will have a diagnosis of sarcoidosis without diabetes, the second group will have a diagnosis of both sarcoidosis and diabetes, and the third group will have a diagnosis of diabetes without sarcoidosis. Sample size is not pre-determined, but investigators anticipate this number to be less than 100. These patients will be asked in person during an office visit to join the study. For each patient who agrees to join, at a clinic visit, investigators will review and sign consent. Following the visit or at a time convenient for each patient, study subjects will undergo a fasting plasma venous sample collection for a hemoglobin A1c, C peptide, insulin level and perform a 2-hour oral glucose tolerance test. The degree of glucose intolerance and prevalence of diabetes will be analyzed and compared between the groups and to historical published control data via T test comparisons. At a later separate visit, patients recruited will undergo ultrasound of the pancreas to assess pancreatic size and morphology.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient referred to or followed in UAB pulmonary clinic with an established diagnosis of sarcoidosis. Any adult patient followed in UAB endocrinology clinic with a diagnosis of diabetes mellitus (excluding type 1 diabetes).

Exclusion Criteria:

* Type 1 diabetes and/or chronic use of corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One group will consist of patients referred to or followed at UAB pulmonary clinic with an established diagnosis of sarcoidosis without diabetes mellitus. A second group will consist of patients referred to or followed at UAB pulmonary and/or endocrinology clinic with diagnoses of both sarcoidosis and diabetes mellitus. A third group will consist of patients referred to or followed at UAB endocrinology clinic with a diagnosis of diabetes mellitus without sarcoidosis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in glucose during oral glucose tolerance test (oGTT) | Baseline

SECONDARY OUTCOMES:
Change in C peptide over oGTT | Baseline
Change in insulin response oGTT | Baseline
Hemoglobin A1c (HbA1c) | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 1 month after publication
Access Criteria: IPD will be shared with future participating researchers who are not yet identified (future fellow physicians).